CLINICAL TRIAL: NCT01153529
Title: CSP #575 - Post-Deployment Afghanistan/Iraq Trauma Related Inventory of Traits (PATRIOT): Phase 1 (Feasibility Study)
Brief Title: Post-Deployment Afghanistan/Iraq Trauma Related Inventory of Traits (PATRIOT): Phase 1 (Feasibility Study)
Acronym: PATRIOT
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 575
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: PTSD
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: OEF/OIF Veterans

SUMMARY:
The long-term goal of this research project is to identify genes that contribute to or guard against developing posttraumatic stress disorder (PTSD) and to better understand how genes and life experiences work together to impact PTSD. Inherited traits are passed down from one generation to the next in genes. Genes contain molecules called DNA, which contain the information that determines our characteristics and carries instructions for constructing and operating our body. Most human diseases have an inherited element. In addition, we, the investigators, hope to learn about how genes and the other materials we find in participants' blood relate to other illnesses and behaviors.

The goal of the feasibility project covered by this application is to test the possibility of conducting research on a large number of veterans in order to look at the association between genes and PTSD. We are inviting 1,000 OEF/OIF veterans to participate, of these, we are anticipating approximately 250 veterans who have served in Afghanistan and/or Iraq to participate in this study. Although 250 participants is our target enrollment, we plan to enroll all veterans included in our initial mailings who desire to participate. We do not anticipate this to exceed 500 individuals. This phase of the study is expected to last about one year. Specific aims are: 1. evaluation of sampling methods and participation rates; 2. field testing of assessment batteries including reliability and validity; and 3. evaluation of the proposed DNA collection and storage procedures.

DETAILED DESCRIPTION:
PURPOSE:

The primary purpose of this feasibility project is to evaluate the feasibility of collecting a case-control cohort of OEF/OIF veterans that is large enough to make possible the identification of genetic variants that affect the risk for PTSD after exposure to traumatic events.

We will also determine if the DNA samples will be of sufficient quality for subsequent analyses.

The primary purpose of the main project which is not covered by this application is to identify genes that affect the risk of developing PTSD.

* RESEARCH QUESTIONS:

  * A.What will be the participation rates for the proposed recruitment strategy?
  * B.How well will the proposed assessment batteries work and are there components that will need to be modified?
  * C.How well will the proposed sampling methods work?
  * D.Will any proposed study procedures need to be changed to make them work better?
* STUDY AIM:

The specific aims have been developed for this feasibility phase of a main study that will have the goal of identifying the most important genes that influence risk and resilience for PTSD and understanding how those genes interact with environmental stressors to cause (or protect from) the clinical disorder.

The feasibility phase protocol presented here is designed to:

* 1.Evaluate sampling methods and participation rates in the proposed populations to determine recruitment feasibility for the main study,
* 2.Develop field experience with proposed assessment batteries and measure reliability and validity to adjust if necessary for the main study,
* 3.Pilot the feasibility of DNA collection, storage and analysis.

After the feasibility phase is complete, a protocol for the main study will be planned and submitted for scientific peer review.

* METHODS:

The OEF/OIF Roster generated by the Defense Manpower Data Center will be used to obtain a list of veterans who have served in at least one of the two theaters of operation since the beginning of the conflict in Iraq and/or Afghanistan. Access to this roster is managed by the VA Environmental Epidemiology Service (EES). This roster currently contains 1,001,463 veterans, of whom 888,454 are male and 475,155 have sought treatment within the VA. Data points abstracted from the roster include, but are not limited to, name, address, SSN, birth date, combat end date, end service date, separation date, military branch, and deployment country. To achieve our target enrollment of 250, 1,000 veterans from the roster will be randomly selected for potential participation. After the sample of 1,000 is randomly drawn, the Cooperative Studies Program Coordinating Center (CSPCC) will mail out letters inviting study participation. We expect the initial 1,000 mailings to yield the following results:

* 300 letters will be non-deliverable for which another address search and re-mail will take place. Nevertheless, it is anticipated that 200 letters will remain undeliverable.
* 800 letters will be deliverable out of which 400 are expected to yield no response after 2 weeks. Second reminder letters will be sent to those potential participants.
* 500 will respond within 2 more weeks with 250 willing to participate (including stated willingness to provide DNA sample) and 250 not interested in participation.

If the above estimates do not yield a minimum of 250 participants, a second wave of mailings will be sent to a new sample of potential participants (N to be determined based on participation rate from the first N = 1000 mailings). Although 250 participants is our target enrollment, we plan to enroll all veterans included in our initial mailings who desire to participate. We do not anticipate this to exceed 500 individuals.

Potential participants will indicate their interest in this study by returning the response letter or by directly calling a dedicated toll-free telephone number. The VA website (http://www.csp.research.va.gov/ ) will have both descriptive information about the study which participants may view at any time as well as the approved informed consent documents. Participants will have an opportunity to ask questions about the study by contacting the study team at CSPCC. The information that we plan on including in the website is as follows:

* DATA SAFETY MONITORING PLAN:

While loss of confidentiality cannot be guaranteed and could be a possible risk, steps will be taken to minimize the risk of loss of confidentiality. First, all collected data received by the Cooperative Studies Program Coordinating Center will be stored in locked file cabinets in a locked office to which only study team members will have access. In addition, Study ID numbers will be used to identify materials with participant responses. Any identifying information will be maintained separately (locked cabinet in a different office).

With regards to participant discomfort, the participants are reminded at the beginning of the interview that they can refuse to answer any questions and discontinue participation at any time. If issues related to trauma memories arise, the participants are asked if they want to be contacted by the study clinician or if they would like to be provided with other medical/mental health resources. Participants will also be asked if they need a break at different intervals during the interview should the participant be experiencing any fatigue due to the duration of the survey. If the participant becomes upset, the study clinician will be contacted by the interviewer. If they simply want to talk to the clinician (per exit interview criteria, then they can as well). If the participant requests assistance without being upset or distressed, they will be provided with information to connect with local resources.

The role of the psychologist will be to collaborate with all study staff, work directly with the study clinician, interface with central IRB and will be the first line resource where decisions need to be made and the first line resource for the coordinating center.

The blood sample will be taken by a certified home health nurse who has experience in minimizing and managing venipuncture side effects.

We propose to minimize potential risks related to genetic samples by never revealing genotype information to participants. No genotypes will become part of the participants' medical records. Participant samples will be coded and the same codes will be used to identify participants in the computer database. The computer files will be password protected. Any hard copies will be maintained in locked filing cabinets in a locked office, and the code book will be locked in a different office. Blood samples sent to Massachusetts Veterans Epidemiology Research and Information Center (MAVERIC) will be placed in secure storage. Although these blood samples will not be banked as part of the CSPG001 - VA Genomic Medicine Program: Specimen Collection and Banking Protocol, they will be processed using their approved established procedures.

* DATA ANALYSIS:

Key Feasibility Outcomes and Resultant Decision Processes

* 1. Participation Rate Evaluation:

  * (a)If fewer than 1 in 10 participants are "cases" (i.e., have current PTSD), then feasibility of the main study is in question, as this would require a sample of over 100,000 screening interviews to achieve the future target sample size of N = 10,000 cases.
  * (b) If fewer than 1 in 4 potential participants agree to participate and follow through to providing a DNA sample, then feasibility is in question, as this would indicate a need for more than 4 times as many contacts in order to achieve sufficient screening interviews to yield the final sample. A participation rate lower than 1 in 4 would also indicate sufficient non-representativeness of the sample that findings could be questioned on the basis of unknowable sample biases.
* 2.Assessment Batteries Evaluation and Reliability :

  * (a)Time to complete the paper-and-pencil and interview measures will be recorded, and some measures may be dropped to minimize participant burden.
  * (b)Psychometric properties of customized measures will be determined, and if unsuitable will be dropped, improved, or substituted. Specific critical measures to be evaluated are:

    * i.)PTSD interview components: Comparison of positive and negative predictive values of the War Related Illness and Injury Study Center Questionnaire (Section IV of the telephone interview)
    * ii.)and the Short-Screening Scale for DSM-IV Posttraumatic Stress Disorder screen. Optimum measures require PPV and NPV > 0.8
    * iii.)MINI interview for lifetime and current PTSD: Validity versus CAPS with kappa > 0.7 for lifetime diagnosis
* 3.If the study's response system to participant psychological distress is needed during this phase, the safety plan will be evaluated
* 4.Determine types and frequency of reported psychological distress to the telephone interview. Ensure suitable emergency response plan available for participants who describe psychological distress (e.g., suicidal ideation) during the telephone interview.

ELIGIBILITY:
Inclusion Criteria:

1.Participant must have served in support of Operation Enduring Freedom or Operation Iraqi Freedom (OEF/OIF) as this is a study relevant to these veterans

Exclusion Criteria:

1. Participants who were unconscious for more than 30 minutes. This may impact event recall
2. Lifetime diagnosis and/or treatment of bipolar disorder or schizophrenia. (NOTE: PTSD in the context of these severe psychiatric disorders is likely to be different from PTSD outside of that context. Excluding subjects with severe psychiatric disorders will increase the homogeneity of the sample and our power to detect genetic effects.)
3. Refusal to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: OEF/OIF Veterans
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Murray B Stein, MD MPH, Study Chair — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- See also: Related Info — http://www.mentalhealth.va.gov/